CLINICAL TRIAL: NCT04771923
Title: Tranexamic Acid Versus Adrenaline for Controlling Iatrogenic Endobronchial Bleeding: a Double Blind, Randomized Controlled Trial
Brief Title: Tranexamic Acid Versus Adrenaline for Controlling Iatrogenic Endobronchial Bleeding
Acronym: TAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Goran Glodić, MD, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8.1-21/20-2; 02/21AG
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Bleeding; Hemoptysis
Keywords: Bronchoscopy; Tranexamic acid; Adrenaline
MeSH Terms: conditions — Hemorrhage; Hemoptysis | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic acid
- Adrenaline (Experimental)
  Interventions: Drug: Adrenaline

INTERVENTIONS:
Drug: Tranexamic acid — Topical instillation of tranexamic acid up to 3x. If bleeding is not controlled patients crossover to adrenaline.
  Arms: Tranexamic acid
Drug: Adrenaline — Topical instillation of adrenaline up to 3x. If bleeding is not controlled patients crossover to tranexamic acid.
  Arms: Adrenaline

SUMMARY:
Endobronchial bleeding is a relatively common complication of diagnostic bronchoscopy. Both tranexamic acid and adrenaline are used topically for the control of endobronchial bleeding. The aim of this study is to compare the efficacy of tranexamic acid with adrenaline in controlling iatrogenic endobronchial bleeding after diagnostic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients with endobronchial bleeding during diagnostic bronchoscopy that was not successfully controlled with cold (4°C) normal saline (3 aliquots of 5ml during 60sec)

Exclusion Criteria:

* Any patient with a contraindication for diagnostic flexible bronchoscopy
* Coagulopathy (PV INR >1.3)
* Thrombocytopenia (<50x10^9) or anemia (hgb <80 g/L)
* Direct oral anticoagulant, low molecular weight heparin or antiplatelet drug therapy
* Thrombophilia, history of pulmonary embolism or deep vein thrombosis
* Contraindication for endobronchial application of adrenaline
* Coronary heart disease, cerebrovascular disease, history of tachyarrhythmia
* Uncontrolled pulmonary hypertension
* Cardiovascular decompensation
* Severe hypoxia (PaO2 <60mmHg, SaO2 <90% with an FiO2 >=60%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of successfully controlled iatrogenic endobronchial bleeding in each arm | Until the end of the individual procedure (bronchoscopy), up to 1 minute after each drug application.
  Bleeding control is assessed by the bronchoscopist by visual confirmation of clot formation.

SECONDARY OUTCOMES:
Number (N) of tranexamic acid/adrenaline applications necessary to control endobronchial bleeding | Until the end of the individual procedure (bronchoscopy), up to 1 minute after each drug application..
  Bleeding control is assessed by the bronchoscopist by visual confirmation of clot formation.
Number (N) of recurrent bleeding episodes after instillation of tranexamic acid/adrenaline | During the first 24 hours immediately after the individual procedure (bronchoscopy).
  Recurrent bleeding episodes and hemoptysis requiring medical and/or bronchoscopic intervention.
Percentage (%) of successfully controlled iatrogenic endobronchial bleeding in each arm in relation to the severity of bleeding. | Until the end of the individual procedure (bronchoscopy), up to 1 minute after each drug application..
  As assessed by the bronchoscopist by visual analogue scale (VAS) 1-10 (1 very mild - 10 very severe).
Percentage (%) of successfully controlled iatrogenic endobronchial bleeding in each arm | Until the end of the individual procedure (bronchoscopy), up to 1 minute after each drug application.
  In different indications and methods (transbronchial lung biopsy, endobronchial biopsy, transbronchial needle aspiration, bronchial brushing).
To compare number (N) of adverse events in each arm | During and up to 1 month after the procedure (bronchoscopy).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Zagreb, Zagreb, Croatia

REFERENCES:
- [Derived] Badovinac S, Glodic G, Sabol I, Dzubur F, Makek MJ, Baricevic D, Korsic M, Popovic F, Srdic D, Samarzija M. Tranexamic Acid vs Adrenaline for Controlling Iatrogenic Bleeding During Flexible Bronchoscopy: A Double-Blind Randomized Controlled Trial. Chest. 2023 Apr;163(4):985-993. doi: 10.1016/j.chest.2022.10.013. Epub 2022 Oct 21. PMID 36273651